CLINICAL TRIAL: NCT04920682
Title: Reversal of Moderate (With the Use of Neostigmine 60 mcg/kg) or Superficial (With the Use of Neostigmine 30 mcg/kg) Neuromuscular Blockade Induced by Cisatracurium. A Prospective, Randomized, Controlled and Doubled Blinded Clinical Trial
Brief Title: Reversal of Moderate or Superficial Neuromuscular Blockade Induced by Cisatracurium
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pontificia Universidade Catolica de Sao Paulo (Other)
Responsible Party: Principal Investigator, Eduardo Toshiyuki Moro, Professor, Pontificia Universidade Catolica de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CAAE 39680120.7.0000.5373
Record Dates: First submitted 2021-04-28; First posted 2021-06-10 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Neostigmine; Neuromuscular Blocking Agents; Muscle Weakness
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled and double-blind clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: For each patient, an opaque envelope will be prepared, sealed and numbered sequentially containing the group to which the patient will be allocated. A list of random numbers generated by computer (www.random.org), in blocks of 1: 1: 1: 1, will be used for this purpose. No collaborator in the operating room, surgeon or anesthesiologist involved in the control of anesthesia and data collection will be aware of the content of the solutions (neostigmine with atropine or saline). An anesthesiologist not involved in the study will be responsible for preparing the solutions:
  * solution 1 (administered when TOF = 3) - neostigmine 60 mcg/kg and atropine 30 mcg/kg diluted with SF until 20 mL (group M); neostigmine 30 mcg/kg and atropine 15 mcg/kg diluted with SF to 20 mL (group N) or 0.9% SF 20 mL (group S)
  * solution 2 (administered when T4 / T1> 0.4) - neostigmine 30 mcg/kg and atropine 15 mcg/kg diluted with SF until 20 mL (group M or N) or SF 0.9% 20 mL (group S)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group M (reversion with moderate neuromuscular blockade) (Active Comparator): Administration of neostigmine 60 mcg/kg and atropine 30 mcg/kg when TOF (Train-of-Four) = 3 and saline when TOF (T4 / T1)> 0.4.
  Interventions: Drug: Reversal of moderate neuromuscular blockade
- Group S (reversion with superficial moderate neuromuscular blockade) (Active Comparator): Administration of 0.9% saline solution (SF) when TOF = 3 and neostigmine 30 mcg/kg and atropine 15 mcg/kg when TOF (T4 / T1)> 0.4.
  Interventions: Drug: Reversal of superficial neuromuscular blockade
- Group N (two-step reversal of neuromuscular blockade) (Active Comparator): Administration of neostigmine 30 mcg/kg and atropine 15 mcg/kg when TOF = 3 and neostigmine 30 mcg/kg and atropine 15 mcg/kg when TOF (T4 / T1)> 0.4 .
  Interventions: Drug: Two-step reversal
- Group P (placebo) (Placebo Comparator): Administration of 0.9% saline solution (SF) when TOF = 3 and when TOF (T4 / T1)> 0.4.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Reversal of moderate neuromuscular blockade — Neostigmine 60 mcg/kg when TOF (Train-of-Four) = 3 and saline when TOF (T4 / T1)> 0.4
  Arms: Group M (reversion with moderate neuromuscular blockade)
Drug: Reversal of superficial neuromuscular blockade — Neostigmine 30 mcg/kg when TOF (T4 / T1)> 0.4
  Arms: Group S (reversion with superficial moderate neuromuscular blockade)
Drug: Two-step reversal — Neostigmine 30 mcg/kg when TOF = 3 and neostigmine 30 mcg/kg when TOF (T4 / T1)> 0.4
  Arms: Group N (two-step reversal of neuromuscular blockade)
Drug: Placebo — 0.9% saline solution (SF) when TOF = 3 and when TOF (T4 / T1)> 0.4
  Arms: Group P (placebo)

SUMMARY:
The administration of acetylcholinesterase inhibiting agents (such as neostigmine) has been used to reverse the muscle paralysis induced by non-depolarizing neuromuscular blocking agents. It is not well known whether there is a difference between the time required for complete reversion of moderate neuromuscular blockade (NMB) after the administration of neostigmine in usual doses when compared to the reversion of superficial NMB with the use of a reduced dose of the same agent (excessive doses of neostigmine administered during superficial blocks may cause paradoxical muscle weakness). The aim of the present study will be to compare, by means of a prospective, randomized, controlled and double-blind clinical trial, the times necessary for the reversion of moderate block with neostigmine 60 mcg / kg or for superficial block to reach values of T4 / T1> 0.9 using neostigmine 30 mcg / kg.

DETAILED DESCRIPTION:
INTRODUCTION One of the most frequent events after performing general anesthesia is the incomplete recovery from NMB. 1 Unfortunately, in addition to the unpleasant and unwanted sensation, post-operative residual muscle weakness can generate potentially more serious problems such as difficulty swallowing, airway obstruction, the occurrence of hypoxemia and pulmonary aspiration. 2,3 Hence, the importance of ensuring a complete reversal of non-depolarizing neuromuscular blocking agents before extubation. Traditionally, the administration of acetylcholinesterase inhibiting agents (such as neostigmine) has been used to reverse the muscle paralysis induced by the use of non-depolarizing neuromuscular blocking agents, but there are limitations related to the antagonism of deep neuromuscular blockade 4,5 or the occurrence of paradoxical effect, when excessive doses of neostigmine are administered during superficial blocks, causing muscle weakness 6,7. In view of this scenario, the need for quantitative assessment of neuromuscular monitoring through the stimulation of peripheral nerves is widely recognized to evaluate NMB reversal.3 During deep NMB [Train-of-Four (TOF) = 0 ; Post-Tetanic Count (PTC)> 1], the administration of neostigmine is likely to be inefficient and its administration is not indicated. In these cases, it would be more prudent to wait for the spontaneous regression of the NMB to less intense levels, when the action of neostigmine becomes more effective and safer.1 Even so, when there is light neuromuscular block (TOF = 4; T4 / T1> 0.4), the use of lower doses of neostigmine should be considered, as there is a risk of inducing paradoxical muscle weakness. 9 It is not well known whether there is a difference between the time required for complete reversion of moderate NMB after the administration of neostigmine in usual doses when compared to the reversion of superficial NMB with the use of a reduced dose of the same agent. The aim of the present study will be to compare, by means of a prospective, randomized, controlled and double-blind clinical trial, the times necessary for the reversion of TOF = 3 (moderate block) to T4 / T1 values> 0.9 (with neostigmine 60 mcg / kg) or for T4 / T1> 0.4 (superficial block) to reach values of T4 / T1> 0.9 (with neostigmine 30 mcg / kg). In addition, the times required for the reversion of TOF = 3 to T4 / T1> 0.4 and TOF = 3 to T4 / T1 = 1 will be evaluated, in addition to the probability of reversing the NMB in less than 10 minutes.

METHODS

After approval by the Research Ethics Committee of School of Medical and Health Sciences, Pontifical Catholic University of São Paulo (Sorocaba, São Paulo - Brazil), patients undergoing general anesthesia for nose and ear surgery at Hospital Santa Lucina will be enrolled to this prospective and randomized clinical trial. Patients aged between 18 and 65 years and physical status according to the American Society of Anesthesiologists I and II will be included. The exclusion criteria will be: (i) refusal to participate in the study; (ii) presence of kidney, liver or neuromuscular disease; (iii) contraindication to the use of any of the drugs used in the study or (iv) body mass index (BMI) ≥ 30. Patients will be randomly divided into four groups according to the moment of NMB reversal and the doses of neostigmine and atropine that will be administered:

* Group M (reversion with moderate NMB): administration of neostigmine 60 mcg/kg and atropine 30 mcg/kg when TOF (Train-of-Four) = 3 and saline when TOF (T4 / T1)> 0.4.
* Group S (reversion with superficial NMB): administration of 0.9% saline solution (SF) when TOF = 3 and neostigmine 30 mcg/kg and atropine 15 mcg/kg when TOF (T4 / T1)> 0.4.
* Group N (two-step reversal): neostigmine 30 mcg/kg and atropine 15 mcg/kg when TOF = 3 and neostigmine 30 mcg/kg and atropine 15 mcg/kg when TOF (T4 / T1)> 0.4 .
* Group C (control): administration of 0.9% saline solution (SF) when TOF = 3 and when TOF (T4 / T1)> 0.4.

For each patient, an opaque envelope will be prepared, sealed and numbered sequentially containing the group to which the patient will be allocated. A list of random numbers generated by computer (www.random.org), in blocks of 1: 1: 1: 1, will be used for this purpose. No collaborator in the operating room, surgeon or anesthesiologist involved in the control of anesthesia and data collection will be aware of the content of the solutions (neostigmine with atropine or saline). An anesthesiologist not involved in the study will be responsible for preparing the solutions:

* solution 1 (administered when TOF = 3) - neostigmine 60 mcg/kg and atropine 30 mcg/kg diluted with SF until 20 mL (group M); neostigmine 30 mcg/kg and atropine 15 mcg/kg diluted with SF to 20 mL (group N) or 0.9% SF 20 mL (group S)
* solution 2 (administered when T4 / T1> 0.4) - neostigmine 30 mcg/kg and atropine 15 mcg/kg diluted with SF until 20 mL (group M or N) or SF 0.9% 20 mL (group S)

Study sequence Anesthesia No patient will receive pre-anesthetic medication. After filling out the consent form and arrival at into the operating room, standard American Society of Anesthesiologists monitors will be applied. A venous access will be obtained in an upper limb contralateral to the NMB monitoring. After pre-oxygenation, anesthesia induction will be performed with 0.5 mcg/kg/min remifentanil for 3 minutes followed by propofol bolus (2.0 mg/kg) and cisatracurium 0.10 mg/kg. Maintenance will be performed with remifentanil (0.3 mcg/ kg/min) and propofol (4 to 6 mg/kg/h). Tracheal intubation will be performed when T1 was less than 5%. The ideal weight will be used to calculate the dose of cisatracurium and neostigmine. Ventilation will be controlled, with the tidal volume and respiratory rate adjusted to maintain PETCO2 between 30 and 40 mmHg. When an inadequate anesthesia plan is suspected (movement, sweating, tachycardia, increase in blood pressure> 10% of pre-induction values), the rate of propofol infusion will be increased and if the adequacy is not sufficient, the rate of infusion of remifentanil. Patients who have a systolic blood pressure decrease greater than 30% or heart rate less than 50 bpm will be treated with ephedrine (10 mg) and atropine (0.5 mg), respectively. Hydration will be performed with 0.9% saline (500 ml in the first 30 minutes and 2 ml / kg / h in the following hours). The central temperature will be maintained above 35 degrees Celsius and the peripheral temperature (tenar eminence of the monitored palm) above 32 degrees Celsius. The reversal of the NMB will be performed when TOF = 3 and / or T4 / T1> 0.4 through the administration of the previously prepared solution.

Monitoring of neuromuscular block The NMB will be monitored by the acceleromyography method (TOF Watch; Schering-Plow) as recommended for use in clinical research. 10 The acceleration transducer will be fixed on the volar side in the distal phalanx of the thumb. The venous access and the BP cuff will be positioned on the arm opposite the limb used to monitor the NMB. After cleaning the skin along the path of the ulnar nerve in the forearm, the electrodes will be positioned at the height of the wrist with a distance between 3 to 6 cm between them. Calibration will be performed after automatically after a 50 Hz tetanic stimulus for 5 seconds. The stimulation (TOF 2 Hz 1.5 seconds, supramaximal stimuli, square wave and duration of 0.2 msec) will be applied every 15 seconds for 2 minutes before the administration of cisatracurium. No additional doses of neuromuscular blockade will be administered. As soon as the third response to TOF is obtained, solution number 1 will be administered and the times between the administration of cisatracurium and TOF = 3 and until this value reaches T4 / T1 = 0.4 will be recorded. At this point, the second solution will be administered and the time until the value of the T4 / T1 ratio reaches a value equal to 0.9 will also be recorded. T1> 0.9. Secondary outcomes will be considered, the probability of reversing the NMB in less than 10 minutes and the time required for the reversion of the moderate NMB (TOF = 3) to T4 / T1 = 1. The sample size will be based on a previous study that determined the need for 12 patients per group to detect with a power of 90% and alpha error of 5% a difference between groups equal to or greater than 1.3 standard deviations.11 Considering the possible losses, 60 patients will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 65 years
* Undergoing general anesthesia for nose and ear surgery
* Physical status according to the American Society of Anesthesiologists I and II

Exclusion Criteria:

* Refusal to participate in the study
* Presence of kidney, liver or neuromuscular disease
* Contraindication to the use of any of the drugs used in the study
* Body mass index (BMI) ≥ 30

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-21 (Actual)

PRIMARY OUTCOMES:
Time necessary for the reversal of moderate blockade using neostigmine 60 mcg / kg or for reversal of superficial blockade using neostigmine 30 mcg / kg | Time from cisatracurium administration until T4 / T1 ratio reaches a value equal to 1.0 assessed up to 2 hours
  Time necessary for the reversion of TOF = 3 (moderate block) to T4 / T1 values 1.0 (with neostigmine 60 mcg / kg) or for T4 / T1> 0.4 (superficial block) to reach values of T4 / T1> 1.0 (with neostigmine 30 mcg / kg)

SECONDARY OUTCOMES:
Probability of reversing the NMB in less than 10 minutes | Time from TOF=3 until T4 / T1 ratio reaches a value equal to 1.0 assessed up to 2 hours
  Probability of reversing moderate blockade (with neostigmine 60 mcg/kg), superficial blockade (with neostigmine 30 mcg/kg) or two-step reversal (neostigmine 15 mcg/kg when NMB is moderate followed by an additional dose of neostigmine 15 mcg/kg when NMB is superficial) when compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo T Moro, MD, Principal Investigator — Pontificia Catholic University of São Paulo
Locations (1):
- Santa Lucina Hospital, Sorocaba, São Paulo, Brazil